CLINICAL TRIAL: NCT04865458
Title: A Phase I Single Arm,Open-label,Multiple Study to Evaluate the Tolerability, Safety, Pharmacokinetics of HEC89736 in Patients With Relapsed or Refractory B-cell Hematologic Malignancies
Brief Title: A Study to Evaluate the Tolerability, Safety, Pharmacokinetics of HEC89736 in Patients With Relapsed or Refractory B-cell Hematologic Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC89736-P-01
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Relapsed or Refractory B-cell Hematologic Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEC89736 treatment (Experimental): HEC89736 tablets,25 mg, 50 mg, 100 mg, 150 mg, 200 mg, QD, 28 days for each cycle
  Interventions: Drug: HEC89736

INTERVENTIONS:
Drug: HEC89736 — HEC89736 tablets QD every 28 days for each cycle

SUMMARY:
Evaluate the safety, pharmacokinetics and efficacy of HEC89736 in patients with Relapsed or Refractory B-cell Hematologic Malignancies

ELIGIBILITY:
Inclusion Criteria:

* Age is over 18 years old
* Histologically or cytologically diagnosed patients with recurrent or refractory B-cell malignancies
* ECOG performance status (PS) 0 ~ 1
* Expected survival of > or = 3 months

Exclusion Criteria:

* The use of PI3Ks as the target of anti-tumor drugs progress (due to intolerance group)
* Received any other anti-cancer treatment within 4 weeks
* Unable to swallow, chronic diarrhea and intestinal obstruction, there are many factors that affect drug use and absorption
* Allergy, or known to have a history of allergy to the drug components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicities evaluated with NCI-CTC AE v5.0 after the first dose | Dosing started until the 28th day
  Incidence of dose limited toxicities and associated dose of HEC89736
Adverse events evaluated by NCI CTCAE 5.0 | From the frst dose to within 30 days after the last dose
  Incidence of adverse events and associated dose of HEC89736

CONTACTS AND LOCATIONS:
Overall Officials: Li Jianyong, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Song Yuqing, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No